CLINICAL TRIAL: NCT05824286
Title: Efficacy and Safety of HbA1c Prediction Model Based on Self-monitoring Blood Glucose in Patients With Type 2 Diabetes
Brief Title: HbA1c Prediction Model in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xianghai Zhou, Prof., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDL2022-30
Record Dates: First submitted 2023-04-09; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Blood Glucose Self-Monitoring; HbA1c Prediction Model; Ridge Regression
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HbA1c prediction model group (Experimental): HbA1c was predicted every month based on self-monitoring blood glucose for patients in HbA1c prediction model group. Study physicians adjusted patients' hypoglycemic therapy based on self-monitoring blood glucose records/glycated albumin and predicted HbA1c every month.
  Interventions: Other: HbA1c prediction
- Conventional treatment group (No Intervention): Study physicians adjusted patients' hypoglycemic therapy based on self-monitoring blood glucose records/glycated albumin, without predicted HbA1c.

INTERVENTIONS:
Other: HbA1c prediction — HbA1c prediction model was developed based on fasting capillary blood glucose and postprandial capillary blood glucose from self-monitoring blood glucose. Since HbA1c was measured once every 3 month, self-monitoring blood glucose records were transferred to predicted HbA1c by prediction model every month.
  Arms: HbA1c prediction model group

SUMMARY:
Patients with type 2 diabetes who have poor blood glucose control are enrolled to evaluate the efficacy and safety of the HbA1c prediction model for adjust the hypoglycemic treatment regimen, compared with the conventional treatment using self-monitoring blood glucose or glycated albumin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Diagnosed with type 2 diabetes mellitus, and the hypoglycemic treatment was not limited; The study physicians judged that the hypoglycemic treatment regimen was stable in nearly 8 weeks;
* Have HbA1c results within 4 weeks, and the range was 7.5-11%;
* Willing and able to conduct self-glucose monitoring;
* Have not participated in any other research program in the past 4 weeks.

Exclusion Criteria:

* Type 1 diabetes mellitus;
* Severe hypoglycemia ≥1 time or fasting C-peptide ≤0.80 ng/mL in the past 6 months;
* Diabetic ketosis in the last 1 week;
* Oral or inhaled corticosteroids for more than 14 days within the last 8 weeks;
* Anemia, recent blood transfusion, hemoglobinopathy (hemoglobinosis and thalassemia), use of erythropoietic drugs, undergoing dialysis;
* Pregnancy or breastfeeding;
* Receiving chemotherapy or radiation therapy;
* Have a severe mental illness and cannot complete the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in measured HbA1c from baseline to 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Change in measured HbA1c from baseline to 12 weeks | 12 weeks
The percentages of participants with HbA1c less than 7.0% at 12 weeks | 12 weeks
The percentages of participants with HbA1c less than 7.0% at 24 weeks | 24 weeks
Change in weight from baseline to 24 weeks | 24 weeks
The rate of severe hypoglycemic events and confirmed hypoglycemic events during the 24 weeks of the study | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Ch, China